CLINICAL TRIAL: NCT06575803
Title: Effect of Repressing of Three Pressable Ceramics With Different Weight Percentage on Patient Satisfaction, Microstructure and Biaxial Flexural Strength
Brief Title: Recycling of Three Pressable Ceramics With Different Weight Percentage
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Faculty of Dental Medicine for Girls (Other Government)
Responsible Party: Principal Investigator, Leena Ashry, Principl investigator leena Asahry(Lashry, Faculty of Dental Medicine for Girls
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CROBR-106-1-E2
Record Dates: First submitted 2024-07-23; First posted 2024-08-28 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Plaque; Patient Satisfaction; Caries, Cervical; Post Operative Pain
Keywords: Repressing; Ips Emax press; celtrapress; lisi press; EDAX; SEM; XRD; Patient satisfaction
MeSH Terms: conditions — Plaque, Amyloid; Patient Satisfaction; Root Caries; Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: clinical performance of single restorations fabricated for the patients from pressed and repressed ceramics
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- crowns constructed from repressed ceramics (Experimental): clinical performance of single restorations fabricated for the patients from pressed and repressed ceramics
  Interventions: Other: clinical measurements and evaluation

INTERVENTIONS:
Other: clinical measurements and evaluation — clinical performance of single restorations fabricated for the patients from pressed and repressed ceramics
  Other Names: clinical measurements

SUMMARY:
Introduction: Green dentistry, is high-technology approach that reduces the environmental impact of dental practices, improper disposal of dental materials wastes results in environmental hazards.

Aim of the study: This studied will be performed o evaluate the effect of repressing of three different types of pressable ceramics, Ips Emax press, Lisi press and Celtra press with different weight percentages on patient satisfaction, mechanical properties, microstructural features and composition of these pressable ceramics.

Materials & Methods:

Seventy five ( N=75) pressable ceramic discs will be constructed ,The samples will be divided to three groups (n=25 each) according to types and composition of pressed and repressed ceramics .Group 1: IPS Emax press .Group 2: Gc Lisipress Group 3: Celtrapress . Each group willbe divided into 5 sub-groups (n=5) according to the weight percentage of newly pressed and repressed ceramics. Subgroup A: 100% new ceramics. Subgroup B: 75% new and 25 % repressed ceramic .Subgroup C: 50% new and 50% repressed ceramics. Subgroup D:25%new and 75% repressed ceramics. Subgroup E: 100% repressed ceramics. Biaxial flexural strength will be measured using universal testing machine. X-ray diffraction will be performed to identify the crystalline phases, and a scanning electron microscope will be used to describe microstructural features. Energy dispersive X-ray analysis will be used to evaluate change in composition Also surface hardness will be evaluated. Patient satisfaction, plaque, cervical caries and marginal discoloration will be evaluated in a follow- up of one year (in vivo part).

DETAILED DESCRIPTION:
Methods:

This study will be divided into two parts: I. In vitro and in vivo studies:

In vitro study

1. Sample size calculation.
2. Sample grouping.
3. Fabrication of the ceramic discs.
4. Testing procedures.
5. Statistical analysis

Sample size estimation and statistical power:

ANOVA test was used according to a previous study by Salem et al (2019) (15), the mean values for the fracture strength ranged from 819.366N to 929.724 according to the weight percentage of the newly pressed and repressed ceramics. G power statistical power analysis program (version 3.1.9.2) will be used for sample size calculation . A total sample size of75 (3groups with 5 subgroups, 5 sample in each sub group) will be sufficient to detect a large effect size of 0.52, with an actual power (1-β error) of 0.95(95%) and a significance level (αerror) 0.05 (5%) for two-sided hypothesis test.

Sample preparation In this study, pressable and repressable ceramic discs will be fabricated. Lost wax technique will be used to manufacture disc-shaped ceramic specimens of three types of pressable ceramic.

Sample grouping:

A total of seventy five (N=75) pressable ceramic discs will be fabricated. The samples will be divided to three groups (n=25 each) according types and composition of pressable ceramics that will be used.

Group 1: IPS emax press (pressed and repressed) (n=25) Group 2: Gc Lisipress (pressed and repressed) (n=25) Group 3: Celtrapress (Pressed and repressed) (n=25) Each group will be divided into 5 sub-groups (n=5) according to the weight percentage of newly pressed and repressed ceramics. Subgroup A: Samples will be 100% new ceramics Subgroup B: Samples will be 75% new and 25 %repressed ceramic Subgroup C: Samples will be 50% new and 50% repressed ceramics Subgroup D: samples will be 25% new and 75% repressed ceramics. Subgroup E: Samples will be100% repressed ceramics. Fabrication of the ceramic discs. 3D printed resin specimens will be sprued and invested in a ring system using phosphate bonded investment .The ring will be then placed in a burnout furnace. Ceramic ingots will be plasticized and pressed in its softened state into the hollow place in the investment ring by means of a plunger. After pressing, the pressed discs and sprues will be weighed to calculate the needed weight of ceramic needed for fabrication of the samples. The sprues will be cut.The ceramic that will be repressed will be placed into the opening at the top surface of the investment mold. Ceramic material will be placed in each pressing cycle according to the desired Wt. % of pressed and repressed ceramics

Laboratory steps:

> Fabrication of pressed and repressed ceramic discs,

1. Construction of resin patterns.
2. Spruing of resin patterns.
3. Investing of resin patterns.
4. Resin elimination.
5. Pressing.
6. Divesting.
7. Finishing and polishing of the discs

Construction of the resin patterns:

A digital design of the disc-shaped specimen; ten millimeters in diameter and one and half millimeter in thickness will be designed by computer-aided design software. The specimen design will be printed by a 3d printer. Seventy-five resin disc specimens will be produced

Spruing of resin patterns:

3d printed resin patterns will be sprued following the manufacturer instructions

Pressing:

1. Ceramic material will placed in each pressing cycle according to the desired Wt. % of pressed and repressed.

   Resin elimination:

   Resin will be eliminated according to manufacturer recommendations; the investment ring was placed in the burn out furnace.

   Divesting:

   The length of the plunger will be marked on the cold investment ring, then The ring will be separated using a separating disc. Finishing and polishing of the discs Ceramic discs will be finished according to the manufacturer's instructions and polished.

   Thermo mechanical aging:

   Ceramic disc specimens will be subjected to thermo-mechanical aging (thermocycling and cyclic loading) using chewing simulator integrated with thermocycling protocol to simulate a total of 6 months of clinical chewing conditions.

   Testing procedure:

   Flexural strength will be measured using universal testing machine. Vicker hardness and fracture toughness will be determined by indentation technique.

   Scanning electron microscope will be used to evaluate microstructure of pressed and repressed ceramics X-ray diffraction will be used to evaluate the crystalline phase. Energy dispersive X-ray analysis (EDAX) will be used to evaluate change in composition of pressed and repressed ceramic.

   Scanning electron microscope will be used to evaluate microstructure of pressed and repressed ceramics In vivo part II. Case presentation for the groups. All the groups and sub-groups in the vitro part will be evaluated as a case presentation study.

   Part (I): In vivo study:

   Following randomized clinical trial rules 1. Ethical considerations. 2. Patient selection. 3. Pre-operative phase. 4. Operative phase. 5. Laboratory steps. 6. Cementation. 7. Clinical evaluation.

   Ethical considerations:

   The study proposal was approved by the Research Ethics Committee (REC) of the Faculty of Dental Medicine for girls, Al-Azhar University, under code: Code of approval P-CR-24-02.

   Patients will be informed about the characteristics and aim of the study and will sign an Informed consent.

   Subject and selection criteria:

   This study will be conducted on the patient who need single crowns attending the outpatient clinic of the Crowns and Bridges department, Faculty of Dental Medicine for Girls, Al-Azhar University.

   This study will be conducted after obtaining the approval of Research Ethic Committee (REC),Faculty of Dental Medicine for Girls, Al-Azhar University.

   The entire patients will be informed about the purpose of investigation, clinical procedures, benefits and hazards of the applied materials and procedure. Before initiation of the procedure a written informed consent will be signed by the patients. Inclusion Criteria
   * Patients requesting single crowns for mandibular posterior teeth.
   * Mandibular posterior teeth that will be prepared to receive single crowns should have adequate crown root ratio, periodontal support, exhibited minimal mobility and adequate tooth preparation length to ensure proper resistance and retention form .
   * Cooperative patients. Exclusion Criteria Patients with severe periodontitis, gingival inflammation, parafunction and poor oral hygiene or high caries activity will be excluded from the present study.

   Pre- operative phase:

   A complete case history including (chief complain, personal data, dental and medical history) will be taken orally from each patient.

   Also, periapical radiograph of abutment tooth and pre-operative clinical examination will be performed for each patient.

   Diagnostic casts of the maxillary and mandibular arches will be obtained after pouring alginate impression.

   Operative phase:

   A. Preparation. B. Secondary impression. C. Samples grouping

   Preparation:

   Clinical procedures will be performed on either vital or endodontically treated molars.

   Secondary impression:

   Impression will be taken for each case using Addition silicone impression material and will be poured with type V dental stone.

   Samples' grouping:

   ▪ Patients will be divided into 3 groups according to types and composition of pressable ceramics that will be used. Group 1: IPS emax press (pressed and repressed) Group 2: Gc Lisipress (pressed and repressed) Group 3: Celtrapress (pressed and repressed) Each group will be divided into 5 sub-groups according to the weight percentage of newly pressed and repressed ceramics. Subgroup A: Samples will be 100% new ceramics Subgroup B: Samples will be 75% new and 25 %repressed ceramic Subgroup C: Samples will be 50% new and 50% repressed ceramics Subgroup D: Samples will be 25% new and 75% repressed ceramics. Subgroup E: Samples will be 100% repressed ceramics.

   Laboratory steps:
   * Fabrication of pressed ceramic crowns, subgroup (A):

     1. Construction of wax patterns. 2. Spruing of wax patterns. 3. Investing of wax patterns. 4. Wax elimination. 5. Pressing. 6. Divesting. 7. Finishing and glazing

   Construction of the wax patterns:

   The wax patterns will be constructed using CAD/CAM system.

   The CAD/CAM system include the following:

   Acquisition unit that consists of:
   1. A desktop computer connected to Dental Scanner.
   2. Exocad computer software that is responsible for designing the restoration, then imports an STL file to the milling machine.

   Milling Machine: Wax discs will be milled.

   Spruing of wax patterns:

   Following the manufacturer instructions, milled wax patterns will be sprued.

   Pressing:

   Ceramic material will placed in each pressing cycle according to the desired Wt. % of pressed and repressed ceramics.

   Wax elimination:

   Wax will be eliminated according to manufacturer recommendations; the investment ring was placed in the burn out furnace.

   Divesting:

   The length of the plunger will be marked on the cold investment ring, then the ring will be separated using a separating disc.

   Finishing and glazing of restorations:

   According to the manufacturer's instructions, all crowns will be finished and glazed.

   Cementation:

   The single crowns will be cemented in patient mouth.

   Clinical evaluation:

   Clinical performance of all crowns of the studied subgroups in terms of: marginal discoloration, color stability, fracture, patient satisfaction, will be evaluated at base line (1week), 3 and 6 months after cementation.

   Clinical evaluation will be performed according to:
   * Modified United States Health Service (USPHS) Ryge Criteria, at base line (1 week), 3, 6 and 12 months after cementation.
   * The presence of plaque will be evaluated using the Loe and Silness plaque index.
   * Clinical examination will be performed using a mirror and sharp explorer, radiograph and photograph.

     * Patient satisfaction will be evaluated using a questionnaire

   The patient satisfaction:

   Patient satisfaction of each subgroup will be assessed by using Visual Analogue Scale (VAS) which is documented chart in the form of satisfied or unsatisfied. A questionnaire will be used to evaluate restorations at baseline (1 week after cementation), 3 and 6 months.

ELIGIBILITY:
Inclusion Criteria:

Patients requesting single crowns for mandibular posterior teeth.

* Mandibular posterior teeth that will be prepared to receive single crowns should have adequate crown root ratio, periodontal support, exhibited minimal mobility and adequate tooth preparation length to ensure proper resistance and retention form .
* Cooperative patients.

Exclusion Criteria:

* Patients with severe periodontitis, gingival inflammation, parafunction and poor oral hygiene or high caries activity will be excluded from the present study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Excellent patient satisfaction, good mechanical properties and microstructure of single crown restorations . | 1 year
  Clinical evaluation will be performed according to:
  - Modified United States Health Service (USPHS) Ryge Criteria, at base line (1 week), 3, 6 and12 months after cementation.
Quality and strength of the restoration and | 1 year
  Modified (USPHS) Ryge criteria system was used to evaluate the quality of all crowns.
  Category Evaluated by Score Criteria Fracture evaluated by Visual inspection with dental explorer Score Alpha (A) No evidence of fracture. Bravo (B) Evidence of fracture Category Evaluated by Score Criteria Fracture evaluated by Visual inspection with dental explorer Score Alpha (A) No evidence of fracture. Bravo (B) Evidence of fracture
Good oral hygiene and patient satisfaction | 1 year
  he presence of plaque will be evaluated using the Loe and Silness plaque index. Score 0= no plaque the tooth surface is clean. Score 1= The tooth surface appears clean ,but dental plaque can be removed from the gingival third with a sharp explorer Score 2= Plaque is visible along the gingival margin to naked eye (moderate accumulation) Score 3=Large amount of plaque in sulcus - Clinical examination will be performed using a mirror and sharp explorer, radiograph and photograph.
  . Patient satisfaction will be evaluated using a questionnaire
  The patient satisfaction:
  Patient satisfaction of each subgroup will be assessed by using Visual Analogue Scale (VAS) which is documented chart in the form of satisfied or unsatisfied. A questionnaire will be used to evaluate restorations at baseline (1 week after cementaton), 3 and 6 months
excellent marginal integrity | 1 year
  Marginal discoloration evaluated by Visual inspection with mirror at 45 degrees angel Score Alpha (A) No discoloration Bravo (B)Superficial staining (removable, usually localized). Charlie (C)Deep staining (not removable, generalized).

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Lina Mohamed Mohamed Abdallah Ali Elashry, Ismailia, Ismalia Old University Street
  - Lina Mohamed Mohamed Abdallah Ali Elashry, Cairo, Ismalia

IPD SHARING:
Plan to Share IPD: No